CLINICAL TRIAL: NCT06402786
Title: Wireless HOME Monitoring of Intracranial (BRAIN) PRESSURE
Brief Title: First-in-human Trial of Home Brain Pressure Measured Using Kitea ICP Sensor, Placed During Hydrocephalus Shunt Surgery.
Acronym: HomeICP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Health Research Council, New Zealand (Other); Auckland City Hospital (Other Government); Kitea Health Ltd (Unknown)
Responsible Party: Principal Investigator, Sarah-Jane Guild, Principal Investigator, University of Auckland, New Zealand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADHB-10040
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hydrocephalus
Keywords: Intracranial Pressure
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Kitea ICP Sensor (Experimental): At the same time as this surgery, the Kitea Sensor will be placed in the brain near the shunt. Participants will be asked to make measurements of their brain pressure at home using the Kitea ICP System for the next 3 months. Aside from the placement of the Kitea Sensor and home measurements of ICP using the Kitea ICP system, all clinical interventions will be standard of care.
  Interventions: Device: Kitea ICP Sensor

INTERVENTIONS:
Device: Kitea ICP Sensor — Kitea ICP Sensor placed in brain during shunt surgery.

SUMMARY:
Patients with hydrocephalus have an abnormal build-up of fluid around the brain and need a tube surgically implanted to drain that fluid. Patients and their caregivers live with the constant fear that the tube will block. Warning symptoms include irritability, headaches and vomiting. Unfortunately, there is no way of telling when fluid build-up is causing a rise in brain pressure and potentially impeding blood flow to the brain (life threatening) except for a brain scan in hospital and possibly hospitalisation.

The investigators want to improve the lives of patients with hydrocephalus. They have developed a tool for parents and caregivers to monitor the pressure in the brain remotely via a sensor placed alongside the drainage tube. The device has been shown to be safe and to give reliable brain pressure readings using a large animal model (sheep). This study is a first-in-human safety study to show it is safe for patient use.

DETAILED DESCRIPTION:
Participants with hydrocephalus who are at risk of repeated bouts of hospitalisation associated with shunt failures and therefore likely to benefit from being able to monitor intracranial pressure will be recruited. 10 adult (>16 years) and 10 children (1-15 years) participants will be recruited in a staggered fashion to allow appropriate evaluation of outcomes. Participants will be recruited when they present to hospital requiring a shunt placement (or revision). At the same time as this surgery, the Kitea Sensor will be placed in the brain near the shunt. Participants will be asked to make measurements of their brain pressure at home using the Kitea ICP System for the next 3 months. Aside from the placement of the Kitea Sensor and home measurements of ICP using the Kitea ICP system, all clinical interventions will be standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a condition requiring cerebral spinal fluid shunting who are undergoing initial shunt placement or shunt revision surgery.
* Adults: Age > 16 years; Children: Age >1 and <15

Exclusion Criteria:

* Adults: Unable to give informed consent
* Paediatric: Failure to obtain assent in a cognitively competent child along with parental consent or parent unable to consent.
* Cortical mantle < 20 mm
* Neurologic or other condition that would prevent compliance with protocol
* Terminal illness with expected survival < 1 year
* Unable to participate in follow-up for 3 months (e.g., travelling overseas for an extended period)
* Underlying medical condition that would make the participant more prone to surgical infections
* Other active implanted medical devices e.g. pacemaker, cochlear implant, implantable cardioverter defibrillator, deep brain stimulation devices
* Participants with conditions likely to require radiation therapy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of device related serious adverse events (Safety of the Kitea ICP Sensor) in the 3 months post-surgery | 3 months
  The primary end point for this study is the proportion of recruited participants who have no safety or tolerability issues in the 3 months post-surgery as assessed by a lack of serious adverse events attributable to the Kitea ICP System or participants requesting device removal.

SECONDARY OUTCOMES:
Incidence of device related serious adverse events (Safety of the Kitea ICP Sensor) in the 6 months post-surgery | 6 months
  The secondary safety end point for this study is the proportion of recruited participants who have no safety or tolerability issues in the 6 months post-surgery as assessed by a lack of serious adverse events attributable to the Kitea ICP System or participants requesting device removal.
Recruitment rate | Through study completion, an average of 1 year
  Proportion of all eligible participants who are enrolled over the study duration.
Data completeness of home ICP recordings using the Kitea ICP system. | 3 months
  Wireless home ICP monitoring will be considered successful if 90% of the attempted ICP measures are able to be obtained.
Participant satisfaction with the requested frequency of making ICP recordings using the Kitea ICP System. | 3 months
  As part of the protocol participants will be asked to make daily ICP measurements using the Kieta ICP system for the first 2 weeks after surgery and then make measurements at least every second day for the remainder of the 3 months. A participant survey at 3 months will collect participant feedback on the perceived burden of making those measurements.

OTHER OUTCOMES:
Number of potentially shunt related clinical events where the Kitea ICP measurements would have provided clinically appropriate ICP values. | 3 months
  The Kitea ICP system will not change shunt performance and the presence of the Kitea Sensor will not stop a shunt failing but it is intended that the ICP values recorded will inform decision making around the whether a shunt is failing or not. In this safety and tolerability study, the ICP values will not be used in clinical decision making. However, as an indication of potential future benefit, any clinical event (defined as the participant seeking clinical care) will be categorised along with the Kitea ICP value associated with that event. This will be presented as a confusion matrix including false and true positives (i.e. shunt failures) and false and true negatives (i.e. false alarms).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah-Jane Guild, PhD, Principal Investigator — The University of Auckland
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No